CLINICAL TRIAL: NCT02954796
Title: Phase 1 Study of SGN-CD352A in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Safety Study of SGN-CD352A for Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN352-001
Record Dates: First submitted 2016-10-28; First posted 2016-11-03 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (Dose Escalation) Cohort -1 - 6 (Experimental): SGN-CD352A will be given intravenously (into a vein; IV) every 28 days at increasing doses.
  Interventions: Drug: SGN-CD352A

INTERVENTIONS:
Drug: SGN-CD352A — On the first day of each 28-day cycle, SGN-CD352A will be given IV. The dose of SGN-CD352A is different in each cohort of the study, with the lowest dose in Cohort -1 (4 mcg/kg) and the highest in Cohort 6 (65 mcg/kg). Patients can only be enrolled into a higher dose level arm if lower doses have proven safe.

SUMMARY:
This study tests the safety of a drug called SGN-CD352A, to find out what its side effects are. SGN-CD352A will be given every 4 weeks to a small group of patients with multiple myeloma.

DETAILED DESCRIPTION:
The study will have 2 parts. In the first part, different doses of SGN-CD352A will be given to different patients (each individual patient will get the same dose for all treatments). The doses will be very low at the start of the trial, and will increase only when the lower dose levels are proven safe.

In the second part of the study, up to 2 dose levels that are both safe and show promising activity against MM will be given to more patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM requiring systemic therapy (per the International Myeloma Working Group [IMWG] ).
* Age 18 years or older.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Life expectancy greater than 3 months.
* Received at least 2 prior lines of therapy for MM including an immunomodulatory drug and a proteasome inhibitor.
* Measurable disease, as defined by at least one of the following: Serum M protein 0.5 g/dL or higher, Urine M protein 200 mg/24 hr or higher, Serum free light chain (SFLC) 10 mg/dL or higher, and Abnormal SFLC ratio.
* Adequate hematologic, renal, and hepatic function
* A negative pregnancy test (for females of childbearing potential).
* Patients must provide written informed consent.

Exclusion Criteria:

* Other invasive malignancy within the past 3 years.
* Active cerebral/meningeal disease related to the underlying malignancy.
* Active Grade 3 or higher infection.
* Known to be positive for HIV or known to have active hepatitis B or C.
* Previous allogeneic stem cell transplant.
* Idiopathic interstitial pneumonia or impaired diffusion capacity of the lung for carbon monoxide (DLCO).
* Cerebrovascular or cardiovascular event, or congestive heart failure within the last 6 months.
* Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Type, incidence, severity, seriousness, and relatedness of adverse events (including laboratory abnormalities) | Through 1 month following last dose.
Incidence of dose-limiting toxicity | During Cycle 1 (Trial Days 1-28)

SECONDARY OUTCOMES:
Overall survival | Up to approximately 3 years
Progression-free survival | Up to approximately 3 years
Duration of objective response | Up to approximately 3 years
Duration of complete response | Up to approximately 3 years
Objective response rate | Up to approximately 3 years
Complete response rate | Up to approximately 3 years
Incidence of antitherapeutic antibodies (ATA) | Up to approximately 3 years
Blood concentrations of SGN-CD352A and metabolites | Up to approximately 3 years

OTHER OUTCOMES:
Exploratory biomarkers of SGN CD352A- mediated pharmacodynamic effects | Up to approximately 3 years
CD352 characterization on malignant plasma cells | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary Campbell, MD, Study Director — Seagen Inc.
Locations (11):
- United States (11):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - Holden Comprehensive Cancer Center / University of Iowa, Iowa City, Iowa
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Charles A. Sammons Cancer Center / Baylor University Medical Center, Dallas, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington